CLINICAL TRIAL: NCT01454310
Title: A Prospective Noninferiority Trial to Compare an Acellular Epithelial Skin Substitute With Autologous Split-thickness Skin Grafts in Deep Partial-thickness Burns
Brief Title: An Acellular Epithelial Skin Substitute in Deep Partial-thickness Burns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Harald Franz Selig, MD, research assistant, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUPRA-VS-STSG-2010
Record Dates: First submitted 2011-10-15; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Wound Healing; Scar Formation
Keywords: Skin substitutes; Split-thickness skin graft; Burn wound; Scar formation; Skin quality
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acellular skin substitute (Experimental)
  Interventions: Device: Wound coverage by acellular skin substitute
- Autologous skin graft (Active Comparator)
  Interventions: Device: Autologous skin

INTERVENTIONS:
Device: Wound coverage by acellular skin substitute — Burn wounds are covered by an acellular skin substitute and remains 10-14 days that peals away in line with re-epithelialisation
  Other Names: Suprathel
  Arms: Acellular skin substitute
Device: Autologous skin — Matched burn wound is covered by autologous skin after tangential excision.
  Arms: Autologous skin graft

SUMMARY:
The purpose of the study is to compare an acellular epithelial skin substitute with autologous split-thickness skin grafts (STSGs) in deep partial-thickness burns. The objective is to evaluate skin quality and scar formation by using subjective and objective burn scar assessments in order to present valuable data for another additional option of wound coverage in deep partial-thickness burns. The investigators hypothesized that the acellular epithelial skin substitute is at least not inferior to autologous skin grafts.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* verified deep partial-thickness burns
* early tangential excision of burn wound (3-5 days after trauma)

Exclusion Criteria:

* Pregnancy
* ABSI-Score >13
* Active tumor or immune-mediated disease
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Time (in days +/- standarddeviation) to complete re-epithelialisation in acellular skin substitue area versus autologous skin | 1 year
  Time to complete re-epithelialisation measured in days after surgery

SECONDARY OUTCOMES:
Skin quality- ratio acellular skin substitute/healthy skin versus ratio autologous skin/healthy skin | 1 year
  Quality of the skin is measured two-fold:
  1. Subjective scar scors: Vancouver Scar Scale, Patient and Observer Scar Scale
  2. Objective scar evaluation by a non-invasive suction device, that measures viscoelastic parameter.

CONTACTS AND LOCATIONS:
Overall Officials: Lars P Kamolz, MD, PhD, MSc, Study Chair — Medical University of Vienna; Maike Keck, MD, Principal Investigator — Medical University of Vienna, Department of Plastic and Reconstructive Surgery
Locations (1):
- Medical University of Vienna, Burn Center, Department of Plastic and Reconstructive Surgery, Vienna, Vienna, Austria

REFERENCES:
- [Background] Uhlig C, Rapp M, Hartmann B, Hierlemann H, Planck H, Dittel KK. Suprathel-an innovative, resorbable skin substitute for the treatment of burn victims. Burns. 2007 Mar;33(2):221-9. doi: 10.1016/j.burns.2006.04.024. Epub 2006 Nov 2. PMID 17084030